CLINICAL TRIAL: NCT06284746
Title: Clinical Efficacy and Safety of Tirelizumab Combined With Chemotherapy in the Treatment of HER-2 Negative Locally Advanced Resectable Gastric Cancer
Brief Title: Tirelizumab Combined With Chemotherapy in the Treatment of HER-2 Negative Locally Advanced Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lin Chen (Other)
Responsible Party: Sponsor-Investigator, Lin Chen, Attending physician, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 301Qiaoz
Record Dates: First submitted 2024-02-21; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Locally Advanced Gastric Carcinoma; HER2 Negative; Efficacy; Safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirelizumab combined with neoadjuvant chemotherapy (Experimental): Four cycles of tirolizumab combined with SOX/XELOX neoadjuvant chemotherapy regimen before surgery, followed by laparoscopic D2 gastric cancer radical surgery, and four cycles of adjuvant chemotherapy after surgery.
  Interventions: Drug: Tirolizumab+SOX/XELOX
- standard chemotherapy (Active Comparator): Four cycles of standard chemotherapy regimen (SOX/XELOX regimen) were administered before and after surgery.
  Interventions: Drug: SOX/XELOX

INTERVENTIONS:
Drug: Tirolizumab+SOX/XELOX — Tirolizumab combined with chemotherapy(SOX/XELOX) regimen. The SOX regimen consists of the drugs Tegilol (S-1) and Oxaliplatin. The XELOX regimen consists of the drugs oxaliplatin and capecitabine.
  Arms: Tirelizumab combined with neoadjuvant chemotherapy
Drug: SOX/XELOX — Simple chemotherapy regimen (SOX/XELOX regimen). The SOX regimen consists of the drugs Tegilol (S-1) and Oxaliplatin. The XELOX regimen consists of the drugs oxaliplatin and capecitabine.
  Arms: standard chemotherapy

SUMMARY:
This study objectively analyzes the safety and survival evaluation of perioperative immunotherapy combined with chemotherapy in locally advanced gastric cancer patients through a prospective randomized controlled trial research method; By comparing the pathological response rate, disease-free survival rate, and incidence of adverse events between the combination therapy and chemotherapy alone group, we aim to verify the efficacy and safety of tirelizumab combined with SOX/XELOX chemotherapy in disease control of locally advanced gastric cancer patients, laying the foundation and providing a basis for large-scale multicenter clinical research.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined this study and signed an informed consent form
* Locally advanced gastric or gastroesophageal junction adenocarcinoma confirmed by pathology or histology as HER-2 negative (cT2-4N+M0 Phase II-III)
* The primary lesion can be surgically removed, and the patient is willing to receive surgical treatment
* There are measurable solid tumors (efficacy evaluation standard: RECIST 1.1)
* Tumor evaluation should be conducted through CT scanning or MRI within 28 days before treatment
* ECOG score 0-1
* Life expectancy ≥ 12 months.

Exclusion Criteria:

* Preoperative imaging examination indicates distant or peritoneal metastasis in patients
* Subjects with any known active autoimmune disease
* Serious cardiovascular disease
* The serum of the subjects tested positive for HIV
* Active hepatitis B (HbsAg positive and HBV-DNA ≥ 10 ^ 3copies/mL) or active hepatitis C (HCV antibody positive and HCV-DNA positive, requiring antiviral treatment at the same time)
* Known subjects with previous allergies to macromolecular protein formulations/monoclonal antibody components, or other contraindications to immunotherapy or chemotherapy
* Have a history of alcohol, drug, or substance abuse
* Individuals with a clear history of neurological or mental disorders, such as epilepsy, dementia, and poor compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) | Less than 20 months
  After neoadjuvant therapy, there were no residual surviving tumor cells in the tumor bed during the pathological remission assessment of postoperative specimens.
Objective Response Rate（ORR） | Less than 20 months
  The proportion of patients whose tumor volume has shrunk to a predetermined value and can maintain the minimum time limit requirement is the sum of complete response (CR) and partial response (PR) ratios, with ORR=CR+PR.

SECONDARY OUTCOMES:
Disease-free survival（DFS） | Less than 20 months
  Time from randomization to disease recurrence or (for any reason) death.
Overall survival（OS） | Less than 20 months
  Time from randomization to death (for any reason)
Major Pathologic Response（MPR） | Less than 20 months
  After preoperative treatment, the number of surviving tumors decreases below the threshold that can affect clinical prognosis.
The incidence of adverse events during treatment | Less than 20 months
  Including adverse reactions related to immunotherapy and postoperative complications. Reflecting safety and tolerability.

CONTACTS AND LOCATIONS:
Locations (1):
- General Surgery Institute, China PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Zheng R, Zhang S, Zeng H, Wang S, Sun K, Chen R, Li L, Wei W, He J. Cancer incidence and mortality in China, 2016. J Natl Cancer Cent. 2022 Feb 27;2(1):1-9. doi: 10.1016/j.jncc.2022.02.002. eCollection 2022 Mar. PMID 39035212
- [Background] 曹毛毛；李贺；孙殿钦；何思怡；雷林；彭绩；陈万青. 2000-2019年中国胃癌流行病学趋势分析. 中华消化外科杂志. 2021;20(01):102-109. doi:10.3760/cma.j.cn115610-20201130-00746
- [Background] Hogner A, Moehler M. Immunotherapy in Gastric Cancer. Curr Oncol. 2022 Mar 2;29(3):1559-1574. doi: 10.3390/curroncol29030131. PMID 35323331
- [Background] Xu J, Jiang H, Pan Y, et al. LBA53 Sintilimab plus chemotherapy (chemo) versus chemo as first-line treatment for advanced gastric or gastroesophageal junction (G/GEJ) adenocarcinoma (ORIENT-16): First results of a randomized, double-blind, phase III study. Ann Oncol. 2021;32:S1331. doi:10.1016/j.annonc.2021.08.2133
- [Background] Emens LA, Middleton G. The interplay of immunotherapy and chemotherapy: harnessing potential synergies. Cancer Immunol Res. 2015 May;3(5):436-43. doi: 10.1158/2326-6066.CIR-15-0064. PMID 25941355
- [Background] Kang YK, Chen LT, Ryu MH, Oh DY, Oh SC, Chung HC, Lee KW, Omori T, Shitara K, Sakuramoto S, Chung IJ, Yamaguchi K, Kato K, Sym SJ, Kadowaki S, Tsuji K, Chen JS, Bai LY, Oh SY, Choda Y, Yasui H, Takeuchi K, Hirashima Y, Hagihara S, Boku N. Nivolumab plus chemotherapy versus placebo plus chemotherapy in patients with HER2-negative, untreated, unresectable advanced or recurrent gastric or gastro-oesophageal junction cancer (ATTRACTION-4): a randomised, multicentre, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2022 Feb;23(2):234-247. doi: 10.1016/S1470-2045(21)00692-6. Epub 2022 Jan 11. PMID 35030335
- [Background] King GT, Sharma P, Davis SL, Jimeno A. Immune and autoimmune-related adverse events associated with immune checkpoint inhibitors in cancer therapy. Drugs Today (Barc). 2018 Feb;54(2):103-122. doi: 10.1358/dot.2018.54.2.2776626. PMID 29637937
- [Background] Myers G. Immune-related adverse events of immune checkpoint inhibitors: a brief review. Curr Oncol. 2018 Oct;25(5):342-347. doi: 10.3747/co.25.4235. Epub 2018 Oct 31. PMID 30464684
- [Background] Haanen JBAG, Carbonnel F, Robert C, Kerr KM, Peters S, Larkin J, Jordan K; ESMO Guidelines Committee. Management of toxicities from immunotherapy: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2017 Jul 1;28(suppl_4):iv119-iv142. doi: 10.1093/annonc/mdx225. No abstract available. PMID 28881921
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338